CLINICAL TRIAL: NCT02852720
Title: Pharmacokinetics of Levobupivacaine and Epinephrine for Transversus Abdominis Plane (TAP) Block for Cesarean Section Postoperative Analgesia
Brief Title: Pharmacokinetics of Levobupivacaine After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Héctor Lacassie, M.D., Pontificia Universidad Catolica de Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 160605003
Record Dates: First submitted 2016-07-27; First posted 2016-08-02 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Pain, Postoperative
Keywords: Pharmacokinetics; levobupivacaine; Pregnancy; Cesarean section; Electrocardiography
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine; Anesthesia, Spinal; High-Energy Shock Waves; Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetics (Experimental): A bilateral TAP block will be performed with 20 ml levobupivacaine 0,25% and epinephrine (5ug/ml). After the blockade, venous blood samples will be taken on predefined times.
  Interventions: Drug: Levobupivacaine; Procedure: Spinal anesthesia; Procedure: Peripheral vein canulation; Procedure: Ultrasonography; Device: Holter

INTERVENTIONS:
Drug: Levobupivacaine — After the block procedure, 2 ml blood samples will be taken in defined times to determine the plasma blood levels of levobupivacaine.
  Other Names: Chirocaine
Procedure: Spinal anesthesia — Spinal anesthesia in the L3-L4 or L4-L5 interspace with hyperbaric bupivacaine 0,75% 1,4 ml plus 20 ug fentanyl to achieve a bilateral anesthetic level of T4 determined by pinprick.
  Other Names: Subarachnoid anesthesia
Procedure: Peripheral vein canulation — An intravenous (18-gauge) catheter will be placed under local anesthesia for co hydration and a second IV catheter for venous sampling
  Other Names: Intravenous catheter
Procedure: Ultrasonography — TAP blocks will be performed using a ultrasound Sonosite M-Turbo US machine (Sonosite Inc, Washington) with an L38x 10-5 megahertz (MHz), 38-mm broadband linear array probe.
  Other Names: Ultrasound
Device: Holter — A portable 12-lead Holter (NorthEast Monitoring®, Boston, USA) will record continuously the electrocardiogram (ECG) after the TAP block, for 24 hrs.
  Other Names: Continuous electrocardiogram

SUMMARY:
Transversus abdominis plane (TAP) block provides effective analgesia and is now a standard of care for analgesia after cesarean section. There is no information on levobupivacaine pharmacokinetics post TAP after pregnancy.

Objective: Generate a pharmacokinetic levobupivacaine model and its effect on the electrocardiogram (ECG).

Method: The investigators will study 12 healthy term pregnant patients, scheduled for elective cesarean section under spinal anesthesia. A bilateral TAP block is performed with 20 ml 0.25% levobupivacaine with epinephrine 5 ug/ml. Sensory block will be assessed at 1-2-6 and 12 hours post puncture. 2 ml of venous blood will be obtained at 2-5-10-30-45-60-90 and 180 minutes. With a Holter machine we will study the effect of levobupivacaine plasma levels and the QTc changes.

Expected results: 1) Plasma levobupivacaine levels; 2) Changes in QTc .

DETAILED DESCRIPTION:
Introduction.

Post cesarean section pain control is a challenging task since it is one of the ten most painful surgeries. Multiple strategies have been proposed for pain control, including neuraxial analgesia, systemic opioids, non-opioid drugs and peripheral nerve blocks, among others.

Transversus abdominal plane (TAP) blocks have been proven to provide effective analgesia when used as part of a multimodal analgesic regimen after abdominal surgery and is becoming a popular technique for post cesarean section analgesia, although recent reports of local anesthesia toxicity have raised concerns about its safety in this population. Currently there is no information on the pharmacokinetics of levobupivacaine of the technique in pregnant patients to guide dosing in a safer way.

Our objective is to generate a pharmacokinetic model to characterize the plasmatic levels of levobupivacaine co-administered with epinephrine and its effect on the ECG, for TAP block in post cesarean section patients.

Methods.

After institutional ethics committee approval and written informed consent, 12 term pregnant patients American Society of Anesthesiologists physical status I or II, scheduled for elective cesarean section were recruited in this prospective, single-blind pharmacokinetic study. Patients were excluded if they had any allergy/sensitivity to local anaesthetic, significant renal or liver dysfunction.

An intravenous (18-gauge) catheter was placed under local anesthesia for co hydration. After the initiation of standard monitoring (continuous electrocardiogram, noninvasive arterial blood pressure, and pulse oximetry), all patients received a spinal anesthesia in the L3-L4 or L4-L5 interspace with hyperbaric bupivacaine 0,75% 1,4 ml plus 20 ug fentanyl to achieve a bilateral anesthetic level of T4 determined by pinprick. After surgery, a TAP block was performed with 20 mL of 0.25% levobupivacaine, with epinephrine 1:200.000 (5 ug/ml) on each side, under ultrasound (US) guidance.

One anesthesiologist experienced in the technique performed all of the TAP blocks using a US Sonosite M-Turbo US machine (Sonosite Inc, Washington) with an L38x 10-5 megahertz (MHz), 38-mm broadband linear array probe. A second anesthesiologist evaluated and approved the US images before administration of the mixture. Blocks were performed with a 21 gauge (G), 110-mm spinal Quincke needle (N. Medical Industries Ltd., Japan) using an in-plane approach.

The extent of sensory blockade of the TAP block to temperature, light touch, and sharp touch was determined using ice, cotton wool, and pinprick, respectively at 1, 2, 6 and 12 hrs post block and the metameric extent of the blockade was recorded. 2 mL venous blood samples were obtained at 2, 5, 10, 30, 45, 60, 90 and 180 minutes after the block. The duration of the blockade was also recorded and symptoms of local anesthetic systemic toxicity were assessed on every control.

Concomitantly we studied the effects of the local anesthetic on myocardial electrical conduction to characterize the pharmacodynamics of TAP block. Briefly, a portable 12-lead Holter (NorthEast Monitoring®, Boston, USA) will record continuously the electrocardiogram (ECG). The information will be stored in an external flash memory card to be analyzed retrospectively with ad hoc software (NorthEast Monitoring®, Boston, USA). We will correlate the eventual changes in the QTc segment with levobupivacaine free plasma levels, which translates the effect of local anesthetics on the heart.

Levobupivacaine Assay.

Levobupivacaine was extracted from plasma using liquid-liquid extraction according to the methods described by Adams et al. The internal standard solution (10 mL of mepivacaine, 30 ug/mL) was added to 0.2 mL of plasma, 100 micro(u)L of sodium hydroxide (2 mol/L solution), and 0.6 mL diethyl ether. The mixture was stirred for 1 minute and centrifuged for 5 minutes at 3000 revolutions/min. Subsequently; the organic phase was transferred to another tube to which 0.25 mL of 0.05 N sulfuric acid was added. The mixture was stirred again for another minute and centrifuged for 5 minutes at 3000 revolutions/min. The aqueous phase was transferred to another tube for subsequent injection. An aliquot of 100 micro(u)L was injected into the high-performance liquid chromatography system. The linearity of the method was evaluated in the range of 0.125 to 10 ug/mL, and 3 concentrations (0.75, 3, and 7.5 ug/mL) were extracted during each protocol as controls.

Knudsen have recently reported the unbound bupivacaine plasma levels thresholds for neurologic symptoms in volunteers of 0,11 ug/ml (SD 0,1 ug/ml). Ikeda et al. found that although there were no differences between the concentrations of bupivacaine and levobupivacaine in plasma, levels of unbound bupivacaine in the cerebral extracellular fluid were significantly higher than levobupivacaine. Consequently, we opted to guide our analysis using bupivacaine pharmacokinetic (PK) data.

Statistical analysis.

Based on the design of relatively frequent sampling planned for each patient and assuming a interindividual variability of 50%, similar to that found in a previous study, which allowed the investigators to characterize the pharmacokinetics of levobupivacaine in 11 healthy volunteers with good accuracy, an estimated number of 12 patients is suitable for the purposes of this study.

Pharmacokinetic Analysis

Population parameter estimations

A one-compartment model with first-order input and elimination was used to describe the time profile of serum levobupivacaine concentrations. Population parameter estimates were calculated using nonlinear mixed effects modelling implemented in the program NONMEM (NONMEM 7.3, Icon Development Solutions, USA). The population parameter variability was modeled in terms of random effect (η) variables. Each variable was assumed to have a mean = 0, and a variance, denoted by ω2, was estimated.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnant patients
* American Society of Anesthesiologists physical status I or II, scheduled for elective cesarean section.

Exclusion Criteria:

* Allergy/sensitivity to the local anaesthetic
* Significant renal or liver dysfunction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Levobupivacaine free plasma levels | 180 minutes
  Plasma levobupivacaine will be assessed at defined timepoints after TAP block

SECONDARY OUTCOMES:
EKG | 12 hours
  Continuous portable EKG monitoring to detect possible EKG changes (QTc segment changes) after TAP block

CONTACTS AND LOCATIONS:
Overall Officials: Hector J Lacassie, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico Universidad Catolica de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardsley H, Gristwood R, Baker H, Watson N, Nimmo W. A comparison of the cardiovascular effects of levobupivacaine and rac-bupivacaine following intravenous administration to healthy volunteers. Br J Clin Pharmacol. 1998 Sep;46(3):245-9. doi: 10.1046/j.1365-2125.1998.00775.x. PMID 9764965
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] Weiss E, Jolly C, Dumoulin JL, Meftah RB, Blanie P, Laloe PA, Tabary N, Fischler M, Le Guen M. Convulsions in 2 patients after bilateral ultrasound-guided transversus abdominis plane blocks for cesarean analgesia. Reg Anesth Pain Med. 2014 May-Jun;39(3):248-51. doi: 10.1097/AAP.0000000000000088. PMID 24682078
- [Background] Corvetto MA, Echevarria GC, De La Fuente N, Mosqueira L, Solari S, Altermatt FR. Comparison of plasma concentrations of levobupivacaine with and without epinephrine for transversus abdominis plane block. Reg Anesth Pain Med. 2012 Nov-Dec;37(6):633-7. doi: 10.1097/AAP.0b013e31826c330a. PMID 23038415
- [Background] Karlsson MO, Sheiner LB. The importance of modeling interoccasion variability in population pharmacokinetic analyses. J Pharmacokinet Biopharm. 1993 Dec;21(6):735-50. doi: 10.1007/BF01113502. PMID 8138894
- [Background] Ikeda Y, Oda Y, Nakamura T, Takahashi R, Miyake W, Hase I, Asada A. Pharmacokinetics of lidocaine, bupivacaine, and levobupivacaine in plasma and brain in awake rats. Anesthesiology. 2010 Jun;112(6):1396-403. doi: 10.1097/ALN.0b013e3181d9cc54. PMID 20460991
- [Derived] Lacassie HJ, Rolle A, Cortinez LI, Solari S, Corvetto MA, Altermatt FR. Pharmacokinetics of levobupivacaine with epinephrine in transversus abdominis plane block for postoperative analgesia after Caesarean section. Br J Anaesth. 2018 Aug;121(2):469-475. doi: 10.1016/j.bja.2018.02.070. PMID 30032887